CLINICAL TRIAL: NCT05617300
Title: Mindfulness-based Dementia Care Partner Program to Reduce Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: A21-117
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2023-12

CONDITIONS: Dementia
Keywords: Caregivers; Mindfulness
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBDC course (Experimental): 8 week MBDC Course including 8 weekly 2 hour classes and a retreat (4 hours). Individual classes will be held virtually via web-based video calls.
  Interventions: Behavioral: Mindfulness-Based Dementia Caregiving

INTERVENTIONS:
Behavioral: Mindfulness-Based Dementia Caregiving — Mindfulness Based Stress Reduction (MBSR) is a standardized program that is both psychoeducation and skills-based, which uses mindfulness meditation practices to help people better cope with their emotions. This study uses a version of MBSR designed specifically for care partners of people living with dementia (PLWD) called Mindfulness Based Dementia Caregiving. Mindfulness Based Dementia Caregiving (MBDC) is a program with 8 weekly 2 hour sessions (plus one extended practice 4 hour retreat) including both formal and informal mindfulness practices, role play, and lectures combined with some dementia-specific education. Participants learn how to incorporate mindfulness practices into day-to-day life to help cope with the challenges and stresses of dementia care.

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and fidelity of implementation of the Mindfulness Based Dementia Care (MBDC) program to reduce depressive symptoms in care partners (CPs) of people living with dementia (PLWD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Self-identify as being an informal CP providing caregiving to a PLWD
* Register for an MBDC course through the Presence Care Website

Exclusion Criteria:

* Previous participation in an MBDC program.
* Does not speak and understand either English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Hanson, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 health care systems in Minnesota, California, and Michigan. Information about the program was shared by clinicians during scheduled visits. Site-specific fliers were posted in public spaces and on institutional websites. A bulk mailing of MBDC fliers targeting non-white/Hispanic Minnesotans with MCI or or dementia was sent. Additionally, a new MBDC instructor was trained recruited an in-person cohort of CPs from her predominately African American Church.
Period: Overall Study
Arm/Group | MBDC Course
Started | 130
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MBDC Course
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (11.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 108
  Male | 19
  Unknown/Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 108
  More than one race | 2
  Unknown or Not Reported | 4
Education [Count of Participants; unit: Participants]
  8th grade or less | 0
  Some high school | 0
  High school diploma or GED | 0
  Technical training or Associate degree | 6
  Some college | 9
  College degree | 42
  Graduate studies | 72
  Unknown or not reported | 1
Occupation [Count of Participants; unit: Participants]
  Employed for wages | 23
  Self-employed | 10
  Out of work for 1 year or more | 5
  Out of work for less than 1 year | 0
  A homemaker | 3
  A student | 2
  Retired | 83
  Unable to work | 2
  Unknown or not reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Participation Rate
Description: Number of the participants who attend the first class of their session. Enrolled is defined as a participant who is assigned to a course. Range [0-124]. A value closer to 124 is indicative of greater feasibility.
Time Frame: Baseline
Population: Includes only participants who attended virtual MBDC program (n=124). Six participants were in live, in person course and not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
Participants | 84

2. Primary Outcome: Completion Rate
Description: Percent of the participants who completed courses. Completion is defined as attending a minimum of 6 of the 9 classes. Range [0-100]. A value closer to 100 is indicative of greater feasibility.
Time Frame: 16 weeks
Population: Includes only participants who attended virtual MBDC program (n=124). Eight participants were in live, in person courses and were not analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
percentage of participants | 94.0

3. Primary Outcome: Questionnaire Specific Response Rate
Description: Completeness of questionnaires given over the course of the study. Completeness is defined percent of complete questionnaires.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of complete questionnaires
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
percentage of complete questionnaires | 96.8 (2.2)

4. Secondary Outcome: Change in Care Partner Burden
Description: Measured using Zarit Burden Interview (ZBI-6). Total of 6 questions scored on a 5 point scale (0-4). The sum of the 6 questions in the total score. Range: 0-24. A higher score is indicative of greater caregiver burden. Change in control period compared to change in intervention period.
Time Frame: baseline, post-course at 8 weeks, follow-up at 20 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
score on a scale
  pre- to post-course | -1.1 [-2 to -0.2]
  pre-course to follow-up | -0.8 [-1.8 to 0.2]

5. Secondary Outcome: Change in Symptoms of Depression
Description: Measured using the Center for Epidemiological Studies Depression Scale (CES-D-10). Total of 10 questions scored on a categorical scale (0-3). The sum of the 10 questions is the total score. Range: 0-30. A total value above 10 is considered to be a sign of depression. A higher score represents a greater degree of depressed mood. Change in control period compared to change in intervention period.
Time Frame: baseline, post-course at 8 weeks, follow-up at 20 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
score on a scale
  pre- to post-course | 0.11 [0.03 to 0.4]
  pre-course to follow-up | 0.09 [0.02 to 0.36]

6. Other Pre Specified Outcome: Change in Self-compassion
Description: Measured using "The State Self-Compassion Scale Short Form." Uses a Likert-type scale ranging from 1 to 5. [Range: 12-60] Higher scores indicates more self compassion.
Time Frame: baseline, post-course at 8 weeks, follow-up at 20 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
score on a scale
  pre- to post-course | 0.4 [0.2 to 0.5]
  pre-course to follow-up | 0.4 [0.2 to 0.6]

7. Other Pre Specified Outcome: Change in Mindful Attention Awareness
Description: Measured using The 5-Item Mindful Attention Awareness Scale - State This is a 5-item scale to indicate at what level they relate to specific experiences, aimed at measuring main characteristics of mindfulness: (scale is 0-"not at all" to 6-"very much"). [Range: 0-30] Higher scores indicate elevated levels of mindfulness expression.
Time Frame: baseline, post-course at 8 weeks, follow-up at 20 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MBDC Course
Number analyzed (Participants) | 124
score on a scale
  pre- to post-course | 0.3 [-0.1 to 0.6]
  pre-course to follow-up | 0.5 [0.2 to 0.9]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Includes only participants who attended virtual MBDC program (n=124). Six participants were in live, in person course and not analyzed.
Arm/Group | MBDC Course
All-Cause Mortality (participants affected / at risk) | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124
Other Adverse Events (participants affected / at risk) | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT05617300/Prot_SAP_000.pdf